CLINICAL TRIAL: NCT01564576
Title: The Influence of the Magnitude of Neuromuscular Blockade on the Surgical Conditions During Laparoscopic Sleeve Gastrectomy
Brief Title: Neuromuscular Blockade and Surgical Conditions
Acronym: Sugamadex
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Haim Berkenstadt, Chairman of Anesthesiology, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-12-9237-HB-CTIL
Record Dates: First submitted 2012-03-15; First posted 2012-03-28 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Morbid Obesity
Keywords: Laparoscopic surgery; Anesthesiology; Neuromuscular blockade
MeSH Terms: conditions — Obesity, Morbid | interventions — Rocuronium; Sugammadex

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional neuromuscular blockade (No Intervention): The dose of rocuronium (medication used for NMB during anesthesia)will be adjusted to maintain a depth of NMB of T1 of 10-20% as assessed by a nerve stimulator. At the end of surgery patients will receive neostigmine 2.5 mg and atropine 1 mg to reverse the effect of rocuronium. Extubation will be performed when train-of-four ratio ≥ 0.9.
  Interventions: Drug: Profound neuromuscular blockade (Rocuronium, Rocuronium bromide, sugammadex, Bridion)
- Profound neuromuscular blockade (Experimental): Rocuronium dose will be adjusted to maintain a depth of NMB of zero response to train of four and a post tetanic count of no more than 10 responses. At the end of surgery patients will receive a single bolus dose of 4 mg/kg sugammadex according to ideal body weight + 40%12. Extubation will be performed when train-of-four ratios ≥ 0.9.
  Interventions: Drug: Profound neuromuscular blockade (Rocuronium, Rocuronium bromide, sugammadex, Bridion)

INTERVENTIONS:
Drug: Profound neuromuscular blockade (Rocuronium, Rocuronium bromide, sugammadex, Bridion) — Rocuronium dose will be adjusted to maintain a depth of NMB of zero response to train of four and a post tetanic count of no more than 10 responses. At the end of surgery patients will receive a single bolus dose of 4 mg/kg sugammadex according to ideal body weight + 40%12. Extubation will be performed when train-of-four ratios ≥ 0.9.
  Other Names: Rocuronium, Rocuronium bromide, sugammadex, Bridion

SUMMARY:
The aim of the present study is to prospectively assess whether deep neuromuscular blockade (NMB) (zero response to train of four and a post tetanic count of no more than 10 responses using a nerve stimulator monitoring) until the end of surgery, followed by sugammadex (bridion®) reversal is superior to the present practice of gradual NMB reduction at the end of surgery followed by neostigmine (Prostigmin®, Vagostigmin®) reversal, in patients undergoing laparoscopic sleeve gastrectomy. The investigators hypothesize that providing deep NMB throughout the procedure creates better conditions for surgery, while reversal of deep NMBwith sugammadex (bridion®) will enable quick and full reversal of relaxation and fewer postoperative respiratory events as compared to neostigmine (Prostigmin®, Vagostigmin®)reversal. Participants will be followed for the duration of hospital stay, an expected average of 7 days.

DETAILED DESCRIPTION:
In laparoscopic bariatric procedures, CO2 is used to insufflate the peritoneal cavity and increase the intra-abdominal pressure for optimal exposure and a suitable operating field. However, the increased intra-abdominal pressure during pneumoperitoneum has profound physiological effects including a reduction in urine output,portal venous flow,respiratory compliance,and cardiac output.

Abdominal muscle relaxation and changes in abdominal wall compliance, produced by the use of anesthetics and muscle relaxants, are important contributors for the achievement of optimal surgical field using minimal abdominal pressure. A practical dilemma is how to maintain good surgical conditions till the end of the operative procedure by deep anesthesia and muscle relaxation on one hand, and to have an awake and spontaneously breathing patient at the end of surgery on the other.

Reversal agents are often used to ensure the reversal of nondepolarizing neuromuscular blockade (NMB). The most widely used is the acetylcholinesterase inhibitor neostigmine (Prostigmin®, Vagostigmin®). However, neostigmine is only partially effective when NMB is deep (less then 1 response using train of four monitoring) and may also be associated with adverse effects, such as cholinergic cardiovascular and gastrointestinal events.Sugammadex (bridion®) is a modified gamma cyclodextrin specifically designed for the reversal of NMB induced by the aminosteroid muscle relaxants including rocuronium bromide (Zemuron®, Esmeron®). Sugammadex (bridion®) acts by encapsulating unbound rocuronium bromide (Zemuron®, Esmeron®)molecules and reducing their concentration at the neuromuscular junction.Studies in surgical patients have shown that sugammadex (bridion®) rapidly and safely reverses rocuronium bromide (Zemuron®, Esmeron®)induced NMB. Unlike acetylcholinesterase inhibitors, sugammadex (bridion®) is also effective in the reversal of deep NMB (no response in train of four monitoring or even no response in post tetanic count monitoring).

Laparoscopic weight reduction surgery requires the appropriate use of muscle relaxation; however, uncertainty remains including indeterminate dosing and unpredictable effect. Additionally, the time to the recovery to a train of four (TOF) ratio of 0.9 in the obese [25.9 (6.7, 13.5-41.0) min] and the overweight groups [14.6 (7.7, 3.3-28.5) min] were significantly longer than that in the normal weight group [6.9 (2.0, 3.0-10.7) min]. Therefore, obese patients are at increased risk for residual muscle relaxation following surgery. Sugammadex (bridion®) has recently been found to reach a peak effect faster than neostigmine(Prostigmin®, Vagostigmin®), in obese patients. In this study, the time to a TOFR ≥ 0.9 was 13 min with 50 μg/kg neostigmine (Prostigmin®, Vagostigmin®)and only 1.7 min with 2 mg/kg sugammadex. Therefore, it appears that sugammadex (bridion®) may more predictably prevent the occurrence of residual muscle relaxation compared to neostigmine (Prostigmin®, Vagostigmin®).

The aim of the present study is to prospectively assess whether deep NMB (zero response to train of four and a post tetanic count of no more than 10 responses using a nerve stimulator monitoring) till the end of surgery, followed by sugammadex (bridion®) reversal is superior to the present practice of gradual NMB reduction at the end of surgery followed by neostigmine (Prostigmin®, Vagostigmin®)reversal, in patients undergoing laparoscopic sleeve gastrectomy. The investigators hypothesize that providing deep NMB throughout the procedure creates better conditions for surgery, while reversal of deep muscle relaxation with sugammadex (bridion®) will enable quick and full reversal of relaxation and fewer postoperative respiratory events as compared to neostigmine (Prostigmin®, Vagostigmin®) reversal. Surgical conditions will be assessed by the surgeons, blinded to the treatment given to the patients, on a 1-4 Likert scale in 5 minutes intervals from abdominal insufflation with gas till the end of surgery (estimated time of 120 minutes). Participants will be followed for respiratory adverse events from admission to the post anesthesia care unit to discharge to the surgical department (continuous measurement of hemoglobin oxygen saturation and respiratory rate for an expected average of 3 hours) and from admission to the surgical department till the time of home discharge (measurement of hemoglobin oxygen saturation and respiratory rate every 6 hours for an expected average of 5 days).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status Class I-III, scheduled to undergo elective sleeve gastrectomy

Exclusion Criteria:

* Neuromuscular disorder affecting NMB
* history of malignant hyperthermia
* significant renal dysfunction
* allergy to medications used during general anesthesia
* concurrent use of medications known to interfere with NMBAs or with sugammadex (antibiotics, anticonvulsants, magnesium salts).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Subjective surgeon feedback on the exposure and surgical field. | From abdominal insufflation with gas till the end of surgery (estimated time of 120 minutes).
  The surgeons blinded to the treatment given to the patients will be asked to assess the quality of the surgical fiels using 1-4 likert scale

SECONDARY OUTCOMES:
Incidence of respiratory adverse events | From admission to the post anesthesia care unit till discharge to the surgical department (expected average of 3 hours) and from admission to the surgical department till the time of home discharge (expected average of 5 days).
  The incidence of respiratory events including- hypoxemia (defined as hemoglobin oxygen saturation lower then 92% while breathing room air), pneumonia (elevated body temperature and findings in chest x-ray), and the need for non invasive or invasive mechanical ventilation; will be assessed continuously during the post anesthesia care unit stay and on 6 hours intervals during the surgical department stay.

CONTACTS AND LOCATIONS:
Overall Officials: Haim Berkenstadt, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Background] Daskalakis M, Scheffel O, Weiner RA. High flow insufflation for the maintenance of the pneumoperitoneum during bariatric surgery. Obes Facts. 2009;2 Suppl 1(Suppl 1):37-40. doi: 10.1159/000198252. Epub 2009 Mar 18. PMID 20124777
- [Background] Matot I, Paskaleva R, Eid L, Cohen K, Khalaileh A, Elazary R, Keidar A. Effect of the volume of fluids administered on intraoperative oliguria in laparoscopic bariatric surgery: a randomized controlled trial. Arch Surg. 2012 Mar;147(3):228-34. doi: 10.1001/archsurg.2011.308. Epub 2011 Nov 21. PMID 22106246
- [Background] Nsadi B, Gilson N, Pire E, Cheramy JP, Pincemail J, Scagnol I, Meurisse M, Defraigne JO, Detry O. Consequences of pneumoperitoneum on liver ischemia during laparoscopic portal triad clamping in a swine model. J Surg Res. 2011 Mar;166(1):e35-43. doi: 10.1016/j.jss.2010.10.033. Epub 2010 Nov 24. PMID 21176920
- [Background] Fahy BG, Barnas GM, Nagle SE, Flowers JL, Njoku MJ, Agarwal M. Changes in lung and chest wall properties with abdominal insufflation of carbon dioxide are immediately reversible. Anesth Analg. 1996 Mar;82(3):501-5. doi: 10.1097/00000539-199603000-00013. PMID 8623951
- [Background] Popescu WM, Bell R, Duffy AJ, Katz KH, Perrino AC Jr. A pilot study of patients with clinically severe obesity undergoing laparoscopic surgery: evidence for impaired cardiac performance. J Cardiothorac Vasc Anesth. 2011 Dec;25(6):943-9. doi: 10.1053/j.jvca.2010.11.012. Epub 2011 Jan 12. PMID 21232976
- [Background] Suy K, Morias K, Cammu G, Hans P, van Duijnhoven WG, Heeringa M, Demeyer I. Effective reversal of moderate rocuronium- or vecuronium-induced neuromuscular block with sugammadex, a selective relaxant binding agent. Anesthesiology. 2007 Feb;106(2):283-8. doi: 10.1097/00000542-200702000-00016. PMID 17264722